CLINICAL TRIAL: NCT05206916
Title: Evaluation of Novel Drug Induced Sleep Endoscopy Procedures in Treating Patients With Obstructive Sleep Apnea Syndrome
Brief Title: New Procedures in Treating Patients With Obstructive Sleep Apnea Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Principal Investigator, Fatma hassanien mohamed, assistent lecturer of chest diseases and tuberculosis, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21-12-22
Record Dates: First submitted 2022-01-12; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- evaluation of cryotherapy as treatment for obstructive sleep apnea patients (Other)
  Interventions: Procedure: cryotherapy

INTERVENTIONS:
Procedure: cryotherapy — Cryotherapy at sites of vibration as origin of snoring and site of collapse for patients with obstructive sleep apnea syndrome

SUMMARY:
Drug-induced sleep endoscopy (DISE) used as diagnostic tool but not yet as a therapeutic procedures to manage the upper airway of snorers and obstructive sleep apnea patients in conditions that mimic natural sleep, there are many aspects that need to be standardized in order to obtain reliable and reproducible information result in cryotherapy at sites of vibration as origin of snoring and site of collapse.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25 - 65 years.
2. Diagnosed with mild, moderate to severe OSA based American Acadmey of Sleep Medicine (AASM) severity Index of apnea hypopnea index (AHI) after Polysomnography (AHI ≥ 5-15 mild, ≥15-30 moderate, ≥30 severe) based on a prior sleep study.
3. BMI is between 28 kg/m2 and 40 kg/m2 at enrollment.
4. Negative result for COVID-19 polymerase chain reaction (RT-PCR) test and absence of clinical symptoms for COVID-19.

Exclusion Criteria:

1. Subjects with a high percentage of central apneas suggesting heart failure.
2. Contraindication to general anesthesia or surgery.
3. Craniofacial abnormality (e.g. retrognathia, micrognathia, etc.) thought to be the primary cause of OSA.
4. Obvious fixed upper airway obstructions (tumors, polyps, nasal obstruction).
5. Tonsil size ≥ +3.
6. Previous surgery within 12 weeks of scheduled procedure performed on the soft tissue of the upper airway (e.g., uvula, soft palate or tonsils).
7. Oral cancer or non-healing oral wounds.
8. Presence of symptoms of influenza-like symptoms.
9. History of surgery affecting the tongue [transoral robotic surgery (TORS), semi-glossectomy, radio-frequency ablation of base of tongue (RFBOT), maxillomandibular advancement (MMA), hypoglossal nerve stimulation (HGNS)].
10. History of radiation therapy to neck or upper respiratory tract
11. Surgical resection for cancer or congenital malformations in the larynx, tongue, or throat (with exception of tonsillectomy and/or adenoidectomy).
12. Clinical evidence of severe chronic obstructive or restrictive pulmonary disease (for example chronic bronchitis, emphysema, pulmonary fibrosis).
13. Active, severe pulmonary vascular disease (for example pulmonary arterial hypertension or pulmonary embolism).
14. Currently receiving treatment for severe cardiac valvular dysfunction, new york heart association (NYHA) Class III or IV heart failure, unstable angina or recent (< 12 month) myocardial infarction or severe cardiac arrhythmias.
15. Subjects with bleeding event, known bleeding diathesis, impaired immunity for any reason, or heart attack or stroke within the last 12 months.
16. Clinical evidence of severe renal failure (Stage 4 or 5) undergoing dialysis or expected to institute dialysis within 12 months.
17. History or current clinical evidence of transient ischaemic attack (TIA) or stroke or muscular dysfunction.
18. Taking medications that in the opinion of the consulting physician may alter consciousness, the pattern of respiration, or sleep architecture, such examples being benzodiazepines, opiates, neuroleptics, prescription stimulants, phenothiazine, or any form of chemical substance abuse.
19. History of dementia or active psychiatric disease that may impact study compliance.
20. Females who are pregnant or females of childbearing age with intention to become pregnant during the study period (≤ 3 months from treatment date).
21. Unable and/or unwilling to comply with study requirements or to provide written informed consent.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
value, side effect and impact of cryotherapy in treatment of patients with obstructive sleep apnea syndrome | polysomnography will done after 2 weeks of intervention
  we use drug induced sleep endoscopy during intervention and use polysomnography before the intervention as diagnostic for cases and after intervention for follow up of cases

IPD SHARING:
Plan to Share IPD: No